CLINICAL TRIAL: NCT03988543
Title: Implementation and Evaluation of an Expanded Bilingual Electronic Symptom Management Program Across a Multi-site, Fully-integrated Comprehensive Cancer Center
Brief Title: Bilingual Electronic Symptom Management Program Across Multi-site, Comprehensive Cancer Center
Acronym: NU IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Medicine (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Cella, Professor and Chair, Department of Medical Social Sciences, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1UM1CA233035-01 (NIH); 1UM1CA233035-01 (NIH)
Record Dates: First submitted 2019-05-08; First posted 2019-06-17 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cancer
Keywords: Curative Intent; Non-curative Intent; Survivorship Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This trial design, in conjunction with our aims and measurement strategy, is consistent with a hybrid Type I effectiveness-implementation trial, which primarily tests the clinical effectiveness of an evidence-based intervention while secondarily documenting and evaluating its implementation. The randomized roll-out implementation trial design is in the same class as the commonly-used stepped wedge trial, but is more practical for real-world application due to lower measurement burden on clinics due to using incomplete wedges. To assess implementation at the level of the clinic, and control for patient-level outcome prior to implementation, we use a pragmatic randomized roll-out implementation trial design with an embedded patient-level randomized group-based comparison.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients will receive current standard care of EHR-integrated symptom monitoring.
- Enhanced Care (Experimental): Patient will receive current standard care of EHR-integrated symptom monitoring, plus patient self-management intervention.
  Interventions: Behavioral: Patient Self-management

INTERVENTIONS:
Behavioral: Patient Self-management — Enhanced care (EC) approach aimed to engage participants actively, and to increase self-efficacy, in the monitoring and managing of their symptoms. After patients complete the current EHR-integrated symptom monitoring, they will receive web-based, patient-centered information to gain knowledge on cancer-related outcomes, improve self-management skills, improve communication skills, and empower them to improve motivation and self-management.
  Other Names: Patient Engagement
  Arms: Enhanced Care

SUMMARY:
Cancer, and cancer treatment, cause many symptoms that can negatively affect quality of life. Despite the development of improved symptom management interventions and several evidence- and consensus-based guidelines, their timely delivery remains uneven in the health care system. Our research center, Northwestern University IMPACT (NU IMPACT), builds upon an electronic health record (EHR)-integrated cancer symptom monitoring and management system, currently deployed by our health care system. We are testing the effectiveness of a system-wide symptom management intervention and the EHR-integrated enhanced care approach, which offers a more personalized symptom monitoring and management experience based on a person's unique needs and language (i.e., English or Spanish).

DETAILED DESCRIPTION:
Using a clinic-level randomized roll-out implementation trial design, we will test the effectiveness of an enhanced care (EC) approach aimed to engage participants actively, and to increase self-efficacy, in the monitoring and managing of their symptoms. The existing EHR-integrated symptom monitoring system will constitute usual care (UC), and added patient engagement and activation features will comprise the EC condition.

Project aims target both patient- and system-level outcomes. Aim 1: Implement a fully-integrated oncology symptom assessment and management program across six clinical units that are part of the NMHC healthcare delivery system; Aim 2: Evaluate the impact of the program by conducting a hybrid Type I effectiveness-implementation trial to evaluate the enhanced care program (EC: symptom monitoring & self-management intervention), relative to usual care (UC) on patient- and system-level outcomes; Aim 3: Identify facilitators and barriers to implementation and disseminate to other health systems. We will enroll an estimated 12,671 participants. To address possible contamination effects within each clinical unit, and allow for unit-level data collection for pre- and post-implementation comparison within and across clinical units, 50% will be enrolled and followed prior to program implementation. The other half will be enrolled post-implementation and will be randomly assigned at a 1:1 ratio (stratified by sex and cancer phase; curative intent, non-curative intent & survivorship) to UC versus EC. Fatigue, pain, anxiety, and depression will be assessed using Patient Reported Outcome Measurement Information System (PROMIS®) computerized adaptive tests (CATs). In addition, we will assess patient clinical outcomes, including healthcare utilization, and cancer treatment delivery outcomes.

ELIGIBILITY:
Inclusion Criteria:

Curative Intent Group:

* ≥ 18 years of age;
* medical chart confirmed diagnosis of a solid or hematological malignancy;
* willingness to be randomized (post-implementation only);
* have initiated primary treatment with curative intent within the past 3 months (i.e., as patients receive surgery, standard- or high-dose chemotherapy, biological therapy, and/or radiotherapy);
* provider confirmed planned treatment and follow-up within the Northwestern Medicine HealthCare (NMHC) hospital and clinics;
* able to read English or Spanish; and
* no evidence of dementia; severe psychopathology (i.e., inpatient psychiatric treatment within past 3-months) or visual or motor impairment that would prevent completion of study procedures.

Non-Curative/Palliative Intent Group:

* ≥ 18 years of age;
* medical chart confirmed diagnosis of advanced or metastatic solid or hematological malignancy;
* willingness to be randomized (post-implementation only);
* undergoing cancer treatment with non-curative/palliative intent (e.g., patients with advanced or metastatic disease who receive chemotherapy, biological therapy, and/or radiotherapy to control or slow advance of their disease);
* provider confirmed planned treatment and follow-up within the NMHC hospital and clinics;
* able to read English or Spanish; and
* no evidence of dementia; severe psychopathology (i.e., inpatient psychiatric treatment within past 3-months) or visual or motor impairment that would prevent completion of study procedures.

Cancer Survivorship Group:

* ≥ 18 years of age;
* medical chart confirmed diagnosis of solid or hematological malignancy within the past 2 years;
* willingness to be randomized (post-implementation only);
* completed active cancer treatment with curative intent, including those who may be receiving maintenance or prophylactic cancer treatment;
* provider confirmed planned follow-up (with or without treatment) within the NMHC e hospital and clinics;
* able to read English or Spanish; and
* no evidence of dementia; severe psychopathology (i.e., inpatient psychiatric treatment within past 3-months) or visual or motor impairment that would prevent completion of study procedures.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4104 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Individual-level change overtime related to cancer and cancer treatment symptoms | Change from baseline adverse symptom severity at 12 months
  Symptom severity will be assessed using Patient-Reported Outcomes Measurement Information System (PROMIS) computer adaptive tests (CATs) related to symptoms of pain, fatigue, depression, anxiety, and physical function. CAT question items are dynamically selected for administration from an item bank based upon the respondent's previous answers. Patient usually completes 4-12 items with a high level of measurement precision for each domain.
Adverse symptom severity related to cancer and cancer treatment | Change from baseline PRO-CTCAE adverse event severity at 12 month
  Adverse symptom severity will be assessed using Patient-Reported Outcomes- Common Terminology for Adverse Events (PRO-CTCAE™) assessment. The PRO-CTCAE questionnaire will ask about nausea, constipation, insomnia, vomiting, shortness of breath, and diarrhea.
Healthcare utilization by participant related to managing their cancer and cancer treatment | Change from baseline healthcare utilization at 12 months
  Participant utilization of healthcare services, such as number of emergency room visits, oncology urgent care visits, unscheduled doctor visits, doctor visits, hospital admissions and length of stay, and supportive care needs to manage their cancer and cancer treatment, will be assessed by electronic health records.
Patient Treatment Delivery Satisfaction | Change from baseline treatment delivery satisfaction at 12 months
  Patient satisfaction of their cancer-related care will be assessed using Consumer Assessment of Healthcare Providers and Systems (CAHPS) Cancer Care survey composite measures.

SECONDARY OUTCOMES:
Patient clinical outcome of cancer recurrence (i.e., cancer has come back) | Cancer recurrance at 12 months
  Cancer recurrence will be assessed by electronic health record diagnosis codes in patients in curative intent and survivorship groups.
Patient clinical outcome of cancer progression (i.e., cancer has becomes worse) | Cancer progression at 12 months
  Cancer progression will be assessed by electronic health records diagnosis codes in curative intent and non-curative intent groups.
Patient clinical outcome of second cancer (i.e., completely new and a different type of cancer than the first one) | Second cancer at 12 months
  Second cancer will be assessed by patient medical record diagnosis codes in curative intent, non-curative intent, and survivorship groups.
Overall Survival (i.e., the time from study randomization until death due to any cause) | Overall survival at 12 months (or end of study)
  Overall survival will be assessed by electronic health records in the curative intent and non-curative intent groups.

CONTACTS AND LOCATIONS:
Overall Officials: David Cella, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

REFERENCES:
- [Derived] Nolla KM, Kuharic M, Lancki N, Walsh-Bailey CL, Flores AM, Garcia SF, Jensen RE, Wang Y, Mai Q, Mercer AM, Smith JD, Psihogios AM, Webster KA, Kircher SM, Franklin PD, Cella D, Yanez BR. Patient Portal Engagement in Oncology: Results From the NU IMPACT Study in a Large Health Care System. JCO Clin Cancer Inform. 2025 Dec;9:e2500178. doi: 10.1200/CCI-25-00178. Epub 2025 Dec 10. PMID 41370780
- [Derived] Smith JD, Bedjeti K, Lancki N, Sloss EA, Merle JL, Kircher S, Coughlin A, Metzger S, Webster KA, O'Connor M, Cahue S, Flores AM, Mai Q, Yanez B, Bass M, Jensen RE, Smith AW, Carroll AJ, Barnard C, George CM, Tsarwhas DG, Richardson K, Penedo FJ, Hemming K, Garcia SF, Scholtens DM, Cella D. Implementation outcomes of a symptom management intervention in ambulatory oncology practices evaluated using a cluster randomized stepped-wedge trial design. Implement Sci. 2025 Dec 2. doi: 10.1186/s13012-025-01475-y. Online ahead of print. PMID 41331816
- [Derived] Kuharic M, Merle JL, Cella D, Mitchell SA, DiMartino L, Ridgeway JL, Dizon DS, Paudel R, Austin JD, Wong SL, Flores AM, Cheville AL, Smith JD; IMPACT Consortium. Psychometric evaluation of the NoMAD instrument in cancer care settings: assessing factorial validity, measurement invariance, and differential item functioning. Implement Sci Commun. 2025 Jun 16;6(1):72. doi: 10.1186/s43058-025-00756-3. PMID 40524282
- [Derived] Cella D, Lancki N, Kuharic M, Yanez B, Bass M, Garcia MG, Webster KA, Smith JD, O'Connor M, Coughlin A, Cahue S, Kircher S, Flores AM, Penedo FJ, Jensen RE, Wilder Smith A, Richardson K, Barnard C, George CM, Tsarwhas DG, Scholtens D, Garcia SF. Web-Based Cancer Symptom Self-Management System: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e258353. doi: 10.1001/jamanetworkopen.2025.8353. PMID 40323601
- [Derived] Cella D, Garcia SF, Cahue S, Smith JD, Yanez B, Scholtens D, Lancki N, Bass M, Kircher S, Flores AM, Jensen RE, Smith AW, Penedo FJ. Implementation and evaluation of an expanded electronic health record-integrated bilingual electronic symptom management program across a multi-site Comprehensive Cancer Center: The NU IMPACT protocol. Contemp Clin Trials. 2023 May;128:107171. doi: 10.1016/j.cct.2023.107171. Epub 2023 Mar 28. PMID 36990275